CLINICAL TRIAL: NCT00998894
Title: A Randomized Effectiveness Trial of Early Hemodynamic Support in Patients Demonstrating a "Triple Low" of Mean-arterial Pressure, End-tidal Anesthetic Concentration, and Bispectral Index
Brief Title: Randomized Trial of Alerts in Patients Demonstrating a "Triple Low"
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, d sessler, Professor & Chair, The Cleveland Clinic
Other Study IDs: 09-453
Record Dates: First submitted 2009-10-19; First posted 2009-10-21 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Low Bispectral Index; Low Mean Arterial Blood Pressure; Low End-tidal Anesthetic Concentration
Keywords: BIS; MAC; MAP

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- decision-support alerts: In patients experiencing a Triple Low (a combination of low MAC, low MAP, and low BIS), a warning alert will be generated for clinicians.
- routine practice: In patients experiencing a Triple Low (a combination of low MAC, low MAP, and low BIS), a warning alert will not be generated for clinicians.

SUMMARY:
The investigators propose to test the theory that smart alarms for the Triple Low State incorporated into a decision support system built into an electronic anesthesia record will prompt clinicians to intervene earlier in situations that would otherwise provoke little concern, and that the alert system will reduce 90-day mortality. Specifically, the investigators will test the hypothesis that providing Triple Low alerts reduces 90-day mortality.

ELIGIBILITY:
Inclusion Criteria:

* Adults presenting for non-cardiac surgery under volatile general anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adults presenting for non-cardiac surgery under volatile general anesthesia
Sampling Method: Probability Sample
Enrollment: 9846 (Actual)
Dates: Start 2009-10; Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
90-day mortality | 90-days

SECONDARY OUTCOMES:
30-day mortality | 30-days
Response to alerts | Intraoperative
  Vasopressor administration within 5 minutes or reduction in volatile anesthetic within 15 minutes of Triple Low onset
Hospital-free days within the initial postoperative month | 30-days

CONTACTS AND LOCATIONS:
Overall Officials: Daniel I Sessler, M.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No